CLINICAL TRIAL: NCT01446302
Title: Metabolic and Inflammatory Responses to Hemodialysis and the Effect of a Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IGFHD2-2011
Record Dates: First submitted 2011-09-29; First posted 2011-10-05 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Kidney Failure, Chronic
Keywords: Dialysis; Protein-energy wasting; Insulin-Like Growth Factor I; Insulin-Like Growth Factor Binding Protein 1; Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Double meal on a HD day (Active Comparator): A standardized meal is served 1 h after start of HD and 1 h after end of HD
  Interventions: Dietary Supplement: Double meal
- Single meal on a HD day (No Intervention): A standardized meal is served 1 h after start of HD. After the meal participants fast for 9 h (6 h after end of HD).
- Single meal on a non-HD day (No Intervention): A standardized meal is served 1 h after study start. After the meal participants fast for 9 h.
- Single meal (healthy controls) (No Intervention): A standardized meal is served 1 h after study start. After the meal participants fast for 9 h.

INTERVENTIONS:
Dietary Supplement: Double meal — A standardized meal is served 1 h after start of HD and 1 h after end of HD.
  Arms: Double meal on a HD day

SUMMARY:
The objective of this study is to characterize the hormonal and inflammatory responses to hemodialysis, and to determine the effect of a meal versus fast on the metabolic changes in the post-dialytic phase.

DETAILED DESCRIPTION:
Studies show that hemodialysis (HD) is a protein catabolic event per se and probably contributes to the high prevalence of protein-energy wasting among HD patients. The muscle catabolic effect of HD is probably caused by loss of amino acids (10-12 grams per dialysis session) and by exacerbation of the inflammatory and hormonal disorders already present. Activation of the immune system during HD has been linked to the contact of blood cells with the dialyzer membrane and to bacterial-derived DNA fragments in the dialysis fluid. An intradialytic increase in interleukin-6 (IL-6) has been shown to correlate with muscle protein catabolism, and because IL-6 continues to increase for 2 hours after HD has ended, there might be a considerable "carry-over effect" to the post-dialytic period. Moreover, HD induces significant changes in the insulin/insulin-like growth factor I (IGF-I) signaling pathways. Plasma insulin is cleared by HD, and the bioactivity of IGF-I is reduced by 50% during a 4-hr maintenance HD due to an up-regulation of IGF-binding protein 1 (IGFBP-1), the only acutely regulated IGFBP.

ELIGIBILITY:
Inclusion criteria:

* > 18 years
* stable maintenance hemodialysis for at least 3 months
* well-functioning arteriovenous shunts with recirculation less than 5%
* informed consent

Exclusion criteria:

* diabetes mellitus
* body mass index below 18.5 or above 30.0 kg/m2
* malnutrition (global assessment score C)
* active malignant disease
* immunosuppressive treatment (including glucocorticoid treatment)
* evidence of an ongoing inflammatory disease (including infection and autoimmune disorders)
* pregnancy

Exclusion criteria during the study:

* myocardial infarction or arrythmia with hemodynamic derangements
* permanent thrombosis in the arteriovenous (AV) shunt
* severe infectious disease
* renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in serum Bioactive IGF-I and IGFBP-1 levels during and after hemodialysis | At 1, 2, 3, 5, 6, 7, 9, and 10 hours after start of hemodialysis
Changes in plasma Interleukin-6 and serum hsCRP levels during and after hemodialysis | At 1, 2, 3, 5, 6, 7, 9, and 10 hours after start of hemodialysis

SECONDARY OUTCOMES:
Pulse wave analysis (augmentation index (AIx)) during and after hemodialysis | At 1, 2, 3, ,4, 5, 6, 7, 8, 9, and 10 hours after start of hemodialysis
Mineral metabolism (including calcium, phosphate, PTH, and FGF-23 levels) during and after hemodialysis | At 1, 2, 3, 5, 6, 7, 9, and 10 hours after start of hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Per Ivarsen, MD, PhD, Study Director — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark; Jan Frystyk, MD,PhD,DMSc, Study Director — Department of Endocrinology and Internal Medicine & Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Denmark; Bente Jespersen, MD, DMSc, Study Director — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark; Jens S Christiansen, MD, DMSc, Study Director — Department of Endocrinology and Internal Medicine & Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Denmark; Else Randers, MD, PhD, Study Director — Department of Nephrology, Viborg Regional Hospital, Denmark; Mark Reinhard, MD, Principal Investigator — Department of Nephrology, Aarhus University Hospital, Skejby, Denmark
Locations (2):
- Denmark (2):
  - Department of Nephrology, Aarhus University Hospital, Skejby, Aarhus N
  - Department of Nephrology, Viborg Regional Hospital, Viborg